CLINICAL TRIAL: NCT06331520
Title: Dexamethasone-sparing Based on Netupitant/Palonosetron(NEPA) With Olanzapine for the Effect of Chemotherapy-induced Nausea and Vomiting in Patients Receiving Highly Emetogenic Chemotherapy: a Randomized Noninferiority III Phase Trial
Brief Title: NEPA Combined With Olanzapine, Dexamethasone-sparing for the Effect of CINV in Patients Receiving HEC Regimens
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Director of Phase I Clinical Trial Department; Professor, Chief physician of oncology department, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Desineo
Record Dates: First submitted 2024-01-29; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Chemotherapy-induced Nausea and Vomiting; Highly Emetogenic Chemotherapy
MeSH Terms: conditions — Vomiting | interventions — netupitant; Palonosetron; netupitant, palosentron drug combination; Olanzapine; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NEO-DXMS GROUP (Active Comparator): NEPA(1 capsule, day1, PO)+ Olanzapine(5mg, day1-4, PO)+ dexamethasone(12mg, day1; 8mg day2-4, PO/IV).
  Interventions: Drug: Netupitant / Palonosetron Oral Capsule [Akynzeo]; Drug: Olanzapine; Drug: Dexamethasone Oral
- HALF-DXMS GROUP (Active Comparator): NEPA(1 capsule, day1, PO)+ Olanzapine(5mg, day1-4, PO)+ dexamethasone(6mg, day1, PO/IV)
  Interventions: Drug: Netupitant / Palonosetron Oral Capsule [Akynzeo]; Drug: Olanzapine; Drug: Dexamethasone Oral
- NEO GROUP (Experimental): NEPA(1 capsule, day1, PO)+ Olanzapine(5mg, day1-4, PO).
  Interventions: Drug: Netupitant / Palonosetron Oral Capsule [Akynzeo]; Drug: Olanzapine

INTERVENTIONS:
Drug: Netupitant / Palonosetron Oral Capsule [Akynzeo] — Akynzeo is the fixed-combination antiemetic comprising netupitant (neurokinin-1 receptor antagonist [NK1 RA]) and palonosetron (5-hydroxytryptamine-3 receptor antagonist [5-HT3 RA]).
Drug: Olanzapine — Olanzapine is an effective antipsychotic drug used in psychiatry to treat psychoses, especially schizophrenia and schizoaffective disorders. It belongs to the 2nd generation antipsychotics, its mechanism of action ranks among multireceptor antagonists (MARTA); it affects the dopamine, serotonin, adrenaline, histamine, and muscarinic systems.
Drug: Dexamethasone Oral — synthetic glucocorticoids
  Arms: HALF-DXMS GROUP; NEO-DXMS GROUP

SUMMARY:
The objective of this Prospective, randomized, non inferiority phase III trial is to confirm the efficacy and saftey of dexamethasone-sparing combined with netupitant/palonostron and olanzapine for the prevention of chemotherapy-induced nausea and vomiting in patients receiving highly emetogenic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥18 years old
2. Patients who receive the high-emetic-risk anticancer agents.
3. Patients who do not take a medicine, for example, 5HT3 receptor antagonists, NK1 receptor antagonists, or research related agents, within 3 weeks prior to enrollment.
4. No nausea or vomiting (grade II or above) within 72 hours before the start of chemotherapy.
5. Subject has Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
6. Subject has a life Expectation of at least 12 weeks.
7. In accordance with the indication of chemotherapy and basic requirements： Peripheral haematology: Hb ≥9.0g/dL; absolute neutrophil count ≥1.5×109/L; Platelet count ≥80×109/L Blood biochemistry: Total bilirubin < 1.25×ULN, ALT and AST ≤ 2.5×ULN; If liver metastasis, ALT and AST < 5×ULN, Creatinine ≤ 1×ULN, basic normal serum electrolyte (Na, Ka, Cl, Ca) Other important organs function normally.
8. Female patients of either non-childbearing potential or child-bearing potential use contraceptive methods throughout the clinical trial.
9. Female patients with child-bearing potential must is negative of pregnancy test.
10. Subjects voluntarily and strictly comply with the research protocol requirements and sign a written informed consent
11. Subjects can independently fill out patient diaries.

Exclusion Criteria:

1. Patients receiving moderate or high emetic radioation therapy within 1 week before chemotherapy or day 1 to 5 after chemotherapy.
2. Within 24 hours after chemotherapy, patients receiving any known or potential antiemetic agents and appearing symptoms vomiting, nausea, or mild nausea symptoms.
3. Scheduled to receive inducer or substrate or strong / moderate inhibitor of cytocrome P450 3A4 (CYP3A4) within 3 weeks prior to day 1.
4. Patients who cannot tolerate chemotherapy drugs.
5. Serious cardiovascular, pulmonary disease, diabetes, mental and other diseases.
6. Pregnant , breastfeeding and woman with child-bearing potential who are unwilling or unable to take effective contraceptive measures.
7. Drug addict or alcohol abuse.
8. Hypocalcemia or any other condition that may cause vomiting.
9. Patients has significant factors that affect the absorption of oral medication, such as chronic diarrhea or obstruction.
10. Subjects has hypersensitivity to netupitant/palonostron capsules or any of its excipients.
11. Scheduled to receive any antiemetic agents within 3 weeks prior to day 1(including but not limited to: neurokin-1 (NK1) receptor antagonist, 5-HT3 receptor antagonists, olanzapine, scopolamine,et al.).
12. Scheduled to receive benzodiazepine, opioid or opioid derivatives (except midazolam, temazepam or triazolam)within 1 week before chemotherapy or day 1 to 5 after chemotherapy.
13. Subjects are currently enrolled in an other clinical study with any other clinical trials, investigational drugs or observational studies within 21 days of baseline.
14. Investigators judged other situations that may affect the progress and results of clinical research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 627 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with complete response (CR) | Within 0-120 hours from the initiation of chemotherapy
  Percentage of patients with complete response (CR) defined defined as no vomiting with no use of rescue therapy

SECONDARY OUTCOMES:
Percentage of Patients With CR (acute and delayed) | From the initiation of chemotherapy infusion(0h)up to beginning of day 6(-120 h)
  Percentage of patients with complete response (CR) defined defined as no vomiting with no use of rescue therapy "Acute"period referred to 0-24 h after the initiation of chemotherapy,"delayed"period referred to 24-120 h.
Percentage of patients with overall complete protection(OCP) | During the acute (within 24 hours post-chemotherapy) and delayed (days 2 thorough 5) phases of chemotherapy
  Percentage of patients with overall complete protection(OCP) defined as no emesis, no rescue medication and able mild nausea(VAS≤25mm).
Percentage of patients with overall total control (OTC) | During 0 ~ 24 hours and 0 ~ 168 hours post-chemotherapy
  Percentage of patients with overall total control (OTC) defined as no emesis, no rescue medication and no nausea(VAS≤5mm).
incidence of adverse events | From initiation of chemotherapy to 168 hours after initiation of chemotherapy
  Adverse event s were graded according to NCI CTCAE v 5.0
quality of life questionnaire | From initiation of chemotherapy to 168 hours after initiation of chemotherapy
  Quality of life(QoL) was evaluated by the Chinese version of the self reported Functional Living Index-Emesis (FLIE) questionnaire by individual patients.